CLINICAL TRIAL: NCT00350155
Title: A 16-Day, Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, Parallel-Group Trial Comparing Lumiracoxib 100mg o.d. With Naproxen 500 mg b.i.d. Plus Omeprazole 20mg o.d. and Placebo in Healthy Volunteers to Investigate on the Safety and Tolerability of Lumiracoxib in the Small Bowel.
Brief Title: Video Capsule Endoscopy to Investigate the Safety and Tolerability of Lumiracoxib in the Small Bowel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCOX189A2425
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Healthy Volunteers
Keywords: Video capsule endoscopy, healthy volunteers, naproxen, omeprazole, lumiracoxib, small bowel
MeSH Terms: interventions — lumiracoxib

INTERVENTIONS:
Drug: Lumiracoxib

SUMMARY:
This study is designed to investigate the potential differences in GI safety and tolerability in the small bowel between lumiracoxib, conventional non-selective NSAID (naproxen) with a proton pump inhibitor (omeprazole), or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects

Exclusion Criteria:

* Evidence of cardiovascular, hepatic, gastrointestinal or renal disorders
* Hereditary problems of galactose intolerance, a severe lactase deficiency or glucose-galactose malabsorption syndrome
* Smokers

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2006-05

PRIMARY OUTCOMES:
Percentage of subjects with one or more small bowel mucosal breaks (with or without hemorrhage) detected by video capsule endoscopy

SECONDARY OUTCOMES:
Total number of small bowel mucosal breaks (with or without hemorrhage) detected by video capsule endoscopy
Percentage of subjects with one or more small bowel lesion detected by video capsule endoscopy
Total number of small bowel lesions detected by video capsule endoscopy
Value of small bowel inflammation (as measured by calprotectin test)
Value of lower GI permeability for lumiracoxib (as measured by differential urinary excretion of sugars)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma AG, Study Chair — Novartis Pharmaceuticals
Locations (2):
- Wiesbaden, Germany
- Nottingham, United Kingdom